CLINICAL TRIAL: NCT01914419
Title: Administration of Oxytocin Via Intramuscular Injection and Intravenous Bolus or Intravenous Infusion in the Third Stage of Labor for Prevention of Postpartum Hemorrhage
Brief Title: Oxytocin Via Intramuscular Injection and Intravenous Bolus or Infusion for Prevention of Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: El Galaa Teaching Hospital (Other); University of Alexandria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3000a
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; Oxytocin; Prevention; Third stage of labor; Hemoglobin; Intravenous; Intramuscular; Bolus
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV infusion (Active Comparator): Oxytocin 10 IU will be administered by IV infusion according to randomization assignment as soon as possible after delivery of the baby.
  Interventions: Drug: Oxytocin
- IV bolus (Active Comparator): Oxytocin 10 IU will be administered by IV bolus according to randomization assignment as soon as possible after delivery of the baby.
  Interventions: Drug: Oxytocin
- IM injection (Active Comparator): Oxytocin 10 IU will be administered by IM injection according to randomization assignment as soon as possible after delivery of the baby.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin

SUMMARY:
The study will evaluate whether prophylactic oxytocin administered in the third stage of labor via intravenous (IV) infusion or IV bolus reduces the rate of postpartum hemorrhage compared to intramuscular (IM) injection.

DETAILED DESCRIPTION:
The study will compare the effect of IV infusion or IV bolus to IM oxytocin administration with respect to mean blood loss and the proportion of women who experience blood loss greater than or equal to 500 ml, women who experience blood loss greater than or equal to 350 ml, side effects, adverse events and change in hemoglobin pre- to post-delivery.

ELIGIBILITY:
Inclusion Criteria:

* All women who present in active labor for a live birth at the study hospital will be considered for participation in the study

Exclusion Criteria:

* Planned or transferred for delivery via Cesarean section
* Administration of a pre-delivery uterotonic to induce or augment labor
* Unable to provide informed consent due to mental impairment, distress during labor or other reason

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4983 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of women with postpartum blood loss equal to or greater than 500 mL | 1 hour after delivery of baby
  Postpartum blood loss equal to or greater than 500 mL as measured in a plastic, calibrated container.

SECONDARY OUTCOMES:
Mean postpartum blood loss | 1 hour after delivery of the baby
  Mean blood loss as measured in a plastic, calibrated container.
Proportion of women with postpartum blood loss equal to or greater than 350 mL | 1 hour after delivery of the baby
  Postpartum blood loss equal to or greater than 500 mL as measured in a plastic, calibrated container.
Proportion of women with postpartum blood loss equal to or greater than 1000 mL | 1 hour after delivery
  Postpartum blood loss equal to or greater than 1000 mL as measured in a plastic, calibrated container.
Mean change in hemoglobin pre-delivery to postpartum | At least 12 hours after removal of IV and within 48 hours of delivery of the baby
  Hemoglobin will be measured in g/dL using the Hemocue machine. Pre-delivery hemoglobin will be taken during labor.
Time to delivery of placenta | Within 1 hour of delivery of the baby
  Time interval in minutes between delivery of the baby and delivery of the placenta
Administration of additional oxytocin, other uterotonics or other interventions such as blood transfusion or hysterectomy | Within 1 hour of delivery of the baby
Side effects 1 hour postpartum | 1 hour after delivery of the baby

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Rasha Dabash, MPH, Principal Investigator — Gynuity Health Projects; Ilana Dzuba, MHS, Principal Investigator — Gynuity Health Projects; Jill Durocher, Principal Investigator — Gynuity Health Projects; Dyanna Charles, MPH, Principal Investigator — Gynuity Health Projects
Locations (2):
- Egypt (2):
  - Shatby Maternity Hospital, Alexandria University, Alexandria
  - El Galaa Teaching Hospital, Cairo

REFERENCES:
- [Derived] Oladapo OT, Okusanya BO, Abalos E, Gallos ID, Papadopoulou A. Intravenous versus intramuscular prophylactic oxytocin for the third stage of labour. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD009332. doi: 10.1002/14651858.CD009332.pub4. PMID 33169839
- [Derived] Charles D, Anger H, Dabash R, Darwish E, Ramadan MC, Mansy A, Salem Y, Dzuba IG, Byrne ME, Breebaart M, Winikoff B. Intramuscular injection, intravenous infusion, and intravenous bolus of oxytocin in the third stage of labor for prevention of postpartum hemorrhage: a three-arm randomized control trial. BMC Pregnancy Childbirth. 2019 Jan 18;19(1):38. doi: 10.1186/s12884-019-2181-2. PMID 30658605